CLINICAL TRIAL: NCT04878094
Title: ARIA II: A Phase III Randomized Controlled Trial of Near-Infrared Angiography During Rectosigmoid Resection and Anastomosis in Women With Ovarian Cancer
Brief Title: A Study of Intra-operative Imaging in Women With Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-202
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma
Keywords: Ovarian cancer; PINPOINT; rectosigmoid resection; anastomosis; 21-202; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A (Active Comparator): Randomized to standard technique and assessment of anastomosis without the use of NIR angiography
  Interventions: Diagnostic Test: Endoscopy
- Arm B (Experimental): Randomized to additional assessment of proximal colonic stump and anastomotic perfusion using NIR angiography
  Interventions: Diagnostic Test: Intravenous Indocyanine Green/ICG injection; Diagnostic Test: PINPOINT endoscopic fluorescence imaging system; Diagnostic Test: Endoscopy

INTERVENTIONS:
Diagnostic Test: Intravenous Indocyanine Green/ICG injection — Intravenous Indocyanine Green/ICG injection will be administered for visualization
  Arms: Arm B
Diagnostic Test: PINPOINT endoscopic fluorescence imaging system — After resection the surgeon will use the PINPOINT imaging system to assess perfusion of the colonic stump. The intervention will again be used following establishment of the anastomosis, however this time via a proctoscope to visualize the proximal and distal ends of the rectosigmoid anastomosis.
  Arms: Arm B
Diagnostic Test: Endoscopy — Standard technique and assessment of anastomosis without the use of NIR angiography

SUMMARY:
The purpose of this study is to find out whether using the PINPOINT imaging system intra-operatively can reduce the risk of anastomotic leaks and other complications after surgery for ovarian cancer, compared with standard intra-operative assessments alone. The PINPOINT endoscopic fluorescence imaging system uses a special camera and a fluorescent (glowing) dye that can evaluate the blood flow of the bowel in real-time. If there is an area that appears concerning, the surgeon can correct the problem during the procedure.

ELIGIBILITY:
Participant Inclusion Criteria

Part 1 (pre-operative):

* 18 years or older
* Diagnosed with primary or recurrent ovarian, fallopian tube, or primary peritoneal cancer
* Scheduled to undergo debulking or cytoreductive surgery
* Suspected need for a low anterior rectosigmoid resection at the time of a debulking procedure
* Enrolled and consented before the operation

Part 2 (intra-operative):

* Completed rectosigmoid resection
* Surgeon plans to perform colorectal anastomosis

Participant Exclusion Criteria

Part 1 (pre-operative):

* Documented history of allergic reaction to ICG
* Not approached for study enrollment before undergoing an unexpected low anterior rectosigmoid resection

Part 2 (intra-operative):

* Did not undergo rectosigmoid resection intraoperatively
* Surgical procedure with rectosigmoid resection for any other type of gynecologic malignancy
* Patient requires permanent colostomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of the risk of 30-day postoperative anastomotic leak at the site of rectosigmoid resection, compared with standard intraoperative assessment alone | 45 days post procedure
  To determine whether the use of NIR angiography assessment of perfusion at the time of rectosigmoid resection in a cohort of patients undergoing surgery for ovarian cancer reduces the risk of 30-day postoperative anastomotic leak at the site of rectosigmoid resection, compared with standard intraoperative assessment alone.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leitao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Jefferson Abington Hospital, Willow Grove, Pennsylvania
  - Houston Methodist Cancer Center (Data Collection Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Leitao MM Jr, Iasonos A, Tomberlin M, Moukarzel LA, Price H, Bennetti G, Ramesh B, Chi DS, Long Roche K, Sonoda Y, Al-Niami A, Mueller JJ, Gardner GJ, Broach V, Jewell EL, Kim S, Feinberg J, Abu-Rustum NR, Zivanovic O. ARIA II: a randomized controlled trial of near-infrared Angiography during RectosIgmoid resection and Anastomosis in women with ovarian cancer. Int J Gynecol Cancer. 2024 Jul 1;34(7):1098-1101. doi: 10.1136/ijgc-2024-005395. PMID 38514101
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org